CLINICAL TRIAL: NCT05760729
Title: Gut-brain Axis: Cognitive Dysfunction and Affective Mood Disorders in Patients With Chronic Inflammatory Bowel Diseases
Brief Title: Cognitive Impairment and Affective Mood Disorders in Patients With IBD
Acronym: COGN-IBD-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Oliviu Florentiu Sarb, Medical doctor, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: 4687/01.10.2021
Record Dates: First submitted 2023-02-23; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Mild Cognitive Impairment; Depression; Anxiety; Stress; Quality of Life
Keywords: inflammatory bowel disease; mild cognitive impairment; depression; quality of life; mild cognitive impairment serum biomarkers
MeSH Terms: conditions — Inflammatory Bowel Diseases; Cognitive Dysfunction; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum samples, 5 ml from each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inflammatory bowel disease patients: It is mandatory to have a certain diagnosis of IBD before the inclusion.
  Interventions: Diagnostic Test: Cognitive testing
- Healthy controls: Patients who have never had the diagnosis of inflammatory bowel disease
  Interventions: Diagnostic Test: Cognitive testing

INTERVENTIONS:
Diagnostic Test: Cognitive testing — Cognitive tests will be carried: MOCA, trail making test, digit symbol substitution, forward and backward digit testing.

SUMMARY:
The aim is to evaluate the presence of mild cognitive impairment (MCI) in patients with inflammatory bowel disease (IBD). This will be done by cognitive tests. Along them, screening for depression, anxiety and stress will be done. A blood sample for determining serum values of homocysteine, protein S100-B, amyloid and BDNF will be stored. Patients will be followed-up for 2 years.

DETAILED DESCRIPTION:
The aim is to evaluate the presence of mild cognitive impairment (MCI) in patients with inflammatory bowel disease (IBD). This will be done by cognitive tests. Along them, screening for depression, anxiety and stress will be done. A blood sample for determining serum values of homocysteine, protein S100-B, amyloid and BDNF will be stored. Patients will be followed-up for 2 years.

Study has 3 phases: inclusion, 1 year visit and 2 year visit. Inclusion: consent signing, checking exclusion and inclusion criteria, cognitive testing, blood sample storing, questionnaires for screening.

1. year visit: cognitive testing.
2. year visit: cognitive testing.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of IBD for IBD group.
2. No diagnosis of IBD for healthy controls group.
3. Obtainment of signed informed consent.

Exclusion Criteria:

1. No consent form signed.
2. Pregnancy.
3. Severe organ insufficiency (cardiac, renal, respiratory, liver).
4. Prior severe head trauma.
5. Neoplasia.
6. Prior neurodegenerative disease.
7. Prior diagnosis of cognitive impairment or dementia.
8. Prior cardiac arrest.
9. Use of B9 and B12 vitamin supplements.
10. Involvement in other clinical trials.
11. Unclear diagnosis.
12. Prior psychiatric disorders.
13. Prior use of neuroleptics.
14. Proven history of familiar Alzheimer disease.
15. Alcohol and drugs abuse.
16. Prior stroke.
17. Prior myocardial infarction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with certain diagnosis of IBD (history, histopathology, biopsy from endoscopy).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Montreal cognitive assessment score (MOCA) | inclusion
  MOCA has 0-30 points
Trail Making Test A (TMT-A) | inclusion
  Scored from 0-100 seconds
Trail Making Test B (TMT-B) | inclusion
  Scored from 0-300 seconds
Digit symbol substitution test | inclusion
  0-90 points
Forward digit span testing | inclusion
  0-16 points
Forward digit span testing | 1 year
  0-16 points
Forward digit span testing | 2 years
  0-16 points
Backward digit span testing | inclusion
  0-14 points
Backward digit span testing | 1 year
  0-14 points
Backward digit span testing | 2 years
  0-14 points
Serum homocysteine | inclusion
  mg/dl
Serum brain derived neurotrophic factor (BDNF) | inclusion
  ug/ml
Serum S100-B protein | inclusion
  ug/ml
Serum amyloid | inclusion
  ug/ml
Montreal cognitive assessment score (MOCA) | 1 year
  MOCA has 0-30 points
Montreal cognitive assessment score (MOCA) | 2 years
  MOCA has 0-30 points

SECONDARY OUTCOMES:
Depression score | inclusion
  0-42 points
Quality of life score | inclusion
  0-100 points for each domain 4 domains:
  * Social relationships
  * Environment
  * Physical health
  * Psychological
Stress score | inclusion
  0-42 points
Anxiety score | inclusion
  0-42 points

CONTACTS AND LOCATIONS:
Locations (3):
- Romania (3):
  - Oliviu Florențiu Sârb, Cluj-Napoca, Cluj
  - Clinica de Hepatologie si Gastroenterologie "Digenio", Cluj-Napoca
  - Spitalul Clinic CF Cluj-Napoca, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarb OF, Vacaras V, Sarb A, Iacobescu M, Tantau AI. Cognitive Dysfunction and Affective Mood Disorder Screening in Patients With Chronic Inflammatory Bowel Disease: Protocol for a Prospective Case-Control Study. JMIR Res Protoc. 2023 Oct 12;12:e50546. doi: 10.2196/50546. PMID 37824197